CLINICAL TRIAL: NCT00107185
Title: Phase I Dose Escalation Study of Autologous Tumor Lysate-Pulsed Dendritic Cell Immunotherapy for Malignant Gliomas in Pediatric Patients
Brief Title: Vaccine Therapy in Treating Young Patients Who Are Undergoing Surgery for Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000420930; UCLA-0410044-01
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2012-08

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood high-grade cerebral astrocytoma; recurrent childhood cerebral astrocytoma; childhood oligodendroglioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine (Experimental)
  Interventions: Biological: therapeutic autologous dendritic cells

INTERVENTIONS:
Biological: therapeutic autologous dendritic cells

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells and tumor cells may help the body build an effective immune response to kill tumor cells. Giving vaccine therapy after surgery may be a more effective treatment for malignant glioma.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating young patients who are undergoing surgery for malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity of adjuvant vaccination with autologous tumor lysate-pulsed dendritic cells after surgical resection in pediatric patients with malignant glioma.
* Determine the maximum tolerated dose of this vaccine in these patients.

Secondary

* Determine, preliminarily, the survival of patients treated with this vaccine.
* Determine, preliminarily, the time to tumor progression in patients treated with this vaccine.
* Determine cellular immune response in patients treated with this vaccine.
* Determine age-dependent differences in response to this vaccine, in terms of immunocompetence, in these patients.

OUTLINE: This is a dose-escalation study.

Patients undergo surgical resection to obtain tumor tissue for production of tumor lysate. Patients then undergo leukapheresis to obtain peripheral blood mononuclear cells (PBMC) for generation of dendritic cells (DC). DC are pulsed with tumor lysate to produce an autologous dendritic cell vaccine. Approximately 10-30 days after leukapheresis, patients receive vaccination with autologous tumor lysate-pulsed dendritic cells intradermally on days 0, 14, and 28 in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed at 2 weeks and then every 2 months for 1 year.

PROJECTED ACCRUAL: A total of 3-18 patients will be accrued for this study within 2-4.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed* WHO grade III or IV malignant glioma of 1 of the following subtypes:
* Anaplastic astrocytoma
* Anaplastic oligodendroglioma
* Glioblastoma multiforme NOTE: *Must be confirmed after surgery
* Newly diagnosed OR recurrent disease
* Bidimensionally measurable disease by contrast-enhancing pre-operative MRI
* Surgically accessible tumor for which surgical resection is indicated at the time of initial pre-operative evaluation
* Must have undergone standard surgery* AND either radiotherapy* or chemoradiotherapy*
* Objective evidence of disease by contrast-enhanced brain MRI after completion of standard therapy NOTE: *Completed after study entry but before assignment to study treatment cohorts
* Age 1 to 18
* Performance status Karnofsky 60-100%
* Hematopoietic

  * Hemoglobin ≥ 10 g/dL
  * Absolute granulocyte count ≥ 1,500/mm^3
  * Platelet count ≥ 100,000/mm^3
* Hepatic

  * SGPT and SGOT ≤ 2 times normal
  * Alkaline phosphatase ≤ 2 times normal
  * Bilirubin ≤ 1.5 mg/dL
  * Hepatitis B and C negative
* Renal

  * BUN ≤ 1.5 times normal OR
  * Creatinine ≤ 1.5 times normal
* Immunologic

  * HIV negative
  * Syphilis negative
* At least 2 weeks since prior radiotherapy and recovered
* Negative pregnancy test
* Fertile patients must use effective contraception
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No chemotherapy during and for 4 weeks* after the final dose of study vaccine
* No corticosteroids for at least 10 days before leukapheresis
* No concurrent corticosteroids
* More than 72 hours since prior systemic antibiotics
* No antihistamines for 5 days before and for 5 days after administration of study vaccine

Exclusion Criteria:

* history of immunodeficiency or autoimmune disease that may be exacerbated by immunotherapy, including any of the following:
* Rheumatoid arthritis
* Systemic lupus erythematosus
* Vasculitis
* Polymyositis
* Dermatomyositis
* Scleroderma
* Multiple sclerosis
* Juvenile-onset insulin-dependent diabetes
* active infection
* fever
* allergy to study reagents
* pregnant or nursing
* other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, localized prostate cancer, or carcinoma in situ of the cervix
* unstable or severe medical or psychiatric condition, as determined by the investigator
* underlying condition that would preclude study participation
* concurrent radiotherapy
* prior organ allograft
* concurrent strong painkillers
* other concurrent immune-suppressing medications
* other concurrent investigational agents
* other adjuvant treatment for 4 weeks* after the final dose of study vaccine NOTE: *Unless there is evidence of tumor progression necessitating additional clinically-indicated treatment; patients requiring treatment due to tumor progression are removed from the study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2005-01; Primary Completion 2009-10 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity of adjuvant vaccination with autologous tumor lysate-pulsed dendritic cells after surgical resection in pediatric patients with malignant glioma. | 1 year

SECONDARY OUTCOMES:
survival | 1 year
  survival with this vaccine

OTHER OUTCOMES:
time to progression | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L. Lasky, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States